CLINICAL TRIAL: NCT01555281
Title: Nelfinavir and Lenalidomide/Dexamethasone in Patients With Progressive Multiple Myeloma That Have Failed Lenalidomide-containing Therapy - A Single Arm Phase I/II Trial
Brief Title: Nelfinavir and Lenalidomide/Dexamethasone in Progressive Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: In connection with the restructuring of SAKK, older ongoing studies were analyzed to determine whether a continuation of the trial would still add value to the data analysis, or whether they do not and could therefore be prematurely terminated.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 39/10; 2010-022035-11 (EudraCT Number); 000001246 (Other: SNCTP)
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Kahler Disease; Lenalidomide; Revlimid; Nelfinavir; Viracept; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Nelfinavir; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir and Lenalidomide/Dexamethasone (Experimental): Phase I: Cycles 1-4 (1 cycle = 28 days) Lenalidomide: 25 mg per day p.o., day 1 to 21 Dexamethasone: 40/20 mg per day p.o., days 1, 8, 15, 22 Nelfinavir: Dose escalation in cohorts of 3 patients
  Phase II: Cycles 1-4 (1 cycle = 28 days) Lenalidomide: 25 mg per day p.o., day 1 to 21 Dexamethasone: 40/20 mg per day p.o., days 1, 8, 15, 22 Nelfinavir: Dose established in phase I twice daily p.o., day 1 to 21
  Interventions: Drug: Nelfinavir; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Nelfinavir — In phase II, the recommended dose of nelfinavir will be administered orally twice daily (in the morning and in the evening) on d1-d21 every 28 days for a maximum of 4 cycles
  Other Names: Viracept
Drug: Lenalidomide — 25 mg of lenalidomide (capsules) will be administered orally daily on d1-d21 every 28 days for a maximum of 4 cycles
  Other Names: Revlimid
Drug: Dexamethasone — 40 mg (for patients <75 years) or 20 mg (for patients ≥75 years) of dexamethasone (tablets) will be administered orally once per day on d1, 8, 15 and 22 every 28 days for a maximum of 4 cycles

SUMMARY:
There is a great need for treatment options in patients with multiple myeloma (MM) after failure of the lenalidomide/dexamethasone regimen as there is no established standard active therapy for these patients.

Combining nelfinavir, a drug targeting both the proteasome and PI3K/Akt pathway, with lenalidomide, may restore lenalidomide-sensitivity to the disease as has been shown in vivo for the PI3K/Akt inhibitor perifosine and the proteasome inhibitor bortezomib.

Patients expected to be included in the trial are heavily pretreated and might not be candidates for further intensive therapies. The combination of nelfinavir with lenalidomide/dexamethasone offers also to these patients an alternative. Preliminary experiences in another SAKK trial with the combination of bortezomib and nelfinavir are positive with few side effects with nelfinavir doses of up to 1875 mg twice daily (bid). For the phase I part of the trial a starting dose of 1250 mg nelfinavir bid was chosen, since the necessary plasma concentration of nelfinavir will not be reached with lower doses.

In case of progression during or after the trial treatment any other lenalidomide- or bortezomib-based chemotherapy combination could be an option for the patient. However, the addition of a chemotherapeutic drug like cyclophosphamide or doxorubicin has known side effects like hematological toxicities, nausea, vomiting and hair loss.

The aim of this trial is to demonstrate that the combination of nelfinavir with lenalidomide/dexamethasone is safe (phase I, dose escalation of nelfinavir) and active (phase II). Patients who do not respond to trial medication will stop trial treatment after 4 months of therapy at the latest.

If the combination of nelfinavir with lenalidomide/dexamethasone should prove to be safe and efficient in treatment of lenalidomide-refractory MM, this would be the first orally available treatment for these patients and establish a new class of drugs (human immunodeficiency virus (HIV) protease inhibitors) as active antineoplastic agents in MM. In addition this would establish the concept of "re-sensitizing" patients to lenalidomide therapy and demonstrate the effect of nelfinavir on proteasomal degradation and Akt phosphorylation in cancer patients in vivo.

DETAILED DESCRIPTION:
Disease background:

MM is a plasma cell tumor. It accounted for an estimated 20,180 new cases of cancer and 11,170 deaths in the United States in 2010. With a prevalence of 23 per 100,000 people, MM is an orphan disease (prevalence <5:10,000). The median age at diagnosis is 60-65 years. Although MM remains incurable, unprecedented gains in survival outcomes have been achieved in the last three decades. Survival has been improved mainly in younger patients below the age of 65 with the advent of high-dose melphalan therapy followed by autologous stem cell transplantation (ASCT). In the last 10 years the introduction of novel therapies, such as thalidomide, lenalidomide and bortezomib have further improved overall survival. However, all patients ultimately relapse and will require salvage therapies.

Therapy background:

The main decision criterion for first-line treatment selection is the patient's eligibility for high-dose chemotherapy with melphalan and subsequent ASCT. Patients who are not eligible for this treatment, due to advanced age, comorbidities or poor performance status, are routinely treated with a combination of melphalan, prednisone and a novel agent such as thalidomide, bortezomib or lenalidomide. Currently, patients will relapse from their first line of therapy at a median of 2-3 years from diagnosis. Achieving a near complete remission and maintaining the residual tumor mass under control is considered as the mainstay in current treatment of MM.

Treatment of relapsed/refractory myeloma is based on double or triple combinations with a novel agent such as lenalidomide or bortezomib with dexamethasone and/or cytotoxic drugs such as alkylators and anthracyclines. The choice of a regimen at relapse depends on the frontline therapy as well as disease- or therapy-related comorbidities. Although patients can achieve long lasting remissions with the novel agents MM remains a chronic disease. Patients will invariably relapse or become refractory to second and later line treatments. Therefore new treatment options for late-line patients are required.

The combination of lenalidomide and bortezomib has been reported to show activity in a subset of lenalidomide and bortezomib double-refractory patients in a phase I/II trial and very recent retrospective data suggest that bortezomib containing regimens may be active in lenalidomide-refractory myeloma patients. There are no approved treatment options for lenalidomide and bortezomib double-refractory patients. Possible therapeutic alternatives such as carfilzomib and pomalidomide are still in clinical development and to date no clinical trials are open in Switzerland. Therefore, treatment options for lenalidomide-refractory patients remain very limited.

Preclinical results in the NCI60 cancer cell line panel show that HIV protease inhibitors such as nelfinavir exhibit a wide spectrum of antitumor activity. They inhibit the proliferation of 60 cancer cell lines derived from nine different tumor types. This is consistent with previous reports demonstrating that HIV protease inhibitors are effective in other diseases like MM and Kaposi sarcoma. Nelfinavir induces cell cycle arrest and apoptosis in tumor cells through inhibition of proteasomal degradation and the PI3K/Akt pathway. Therefore preclinical evidence underscores the proteasome inhibiting activity of nelfinavir. Modulation of proteasome function is a rational approach to overcome chemo-resistance and achieve chemo-sensitization, suggesting that the addition of such an agent to myeloma standard treatment could restore sensitivity to the standard therapy.

Pharmacologic intervention with the PI3K/Akt pathway induced cell death in MM cell lines and primary tumor samples. Inhibition of Akt phosphorylation by perifosine has shown significant clinical activity and manageable toxicity in patients with relapsed/refractory MM in combination with dexamethasone alone (≥MR (minor response) of 38%; SD (stable disease) of 47%), or together with both lenalidomide and dexamethasone (≥PR (partial response) of 50%, MR of 20%). These data suggest an important role of the Akt pathway for malignant growth and survival of MM cells also in vivo. The addition of nelfinavir to standard lenalidomide/dexamethasone treatment in lenalidomide-refractory patients is expected to restore sensitivity of the myeloma cells to lenalidomide, acting via inhibition of the PI3K/Akt pathway and modulation of proteasome function.

Aim of this study is to demonstrate the safety and activity of combining lenalidomide and dexamethasone with nelfinavir in patients with progressive MM that have failed lenalidomide-containing therapy.

Treatment Nelfinavir:

Nelfinavir mesylate (Viracept) is an inhibitor of the HIV protease 1. Inhibition of this viral protease prevents cleavage of the Gag and Gag-Pol polyproteins resulting in the production of immature, non-infectious virus. The pharmacokinetic properties of nelfinavir were evaluated in healthy volunteers and HIV-infected patients. No substantial differences were observed between the two groups. In Switzerland the registered dose of nelfinavir for the treatment of HIV-1 infection in combination with other antiretroviral agents is 1250 mg bid or 750 mg three times daily (tid).

Plasma concentrations from a pharmacokinetic study with 10 HIV-positive patients after multiple dosing with 1250 mg twice daily for 28 days were 4.0 mg/L (peak plasma level) and 2.2 mg/L / 0.7 mg/L (morning/evening trough), respectively. Peak plasma concentrations were approximately 6 microM. Nelfinavir in serum is extensively protein-bound (>98%). The area under the curve (AUC) is 1.5 times higher with the bid regimen compared to the tid regimen, without significantly elevated toxicity. The maximal concentration of nelfinavir is usually achieved 3 to 4 hours after administration with food. The effective half-life in blood plasma ranges from 3 to 5 hours. Multi-dose pharmacokinetics of nelfinavir, have not been studied in HIV-positive patients with hepatic or renal insufficiency.

Nelfinavir is an inhibitor of cytochrome P450 3A4 (CYP3A4) and is mainly metabolized by CYP3A4 and CYP2C19. The main metabolite of nelfinavir (the hydroxylated metabolite nelfinavir M8) is also active against HIV and circulates in the plasma at around 30% of the present nelfinavir amount.

The dose limiting toxicity (DLT) has not been defined yet. A respective dose finding trial for nelfinavir mono-therapy in patients with solid tumors is ongoing. Preliminary data from that trial shows that nelfinavir is well tolerated at 2.5 times (2 x 3125 mg/day) the American Food and Drug Administration approved dose for the treatment of HIV infections of 2 x 1250 mg/day with no grade 4-5 clinical toxicities. The most prevalent laboratory abnormalities grade 4 with a dose level (DL) of 3125 mg bid were transaminitis, hyperglycemia and diarrhea. The AUC of nelfinavir in plasma showed a plateau at doses of 1875 mg bid.

A phase I study of Nelfinavir in liposarcoma with a maximum DL of 4250 mg bid shows a peak plasma level of 6.3 mg/L. One patient experienced transient grade 3 pancreatitis after one week of nelfinavir. No other DLTs were observed.

Recent testing of this nelfinavir dose in combination with radiation therapy and weekly gemcitabine (200-300 mg/m2) in patients with pancreatic cancer did not cause increased toxicity in this trial.

The main side effects of nelfinavir include diarrhea (>10%), rash, elevated liver enzymes, and reduced blood counts (1-10%) at the therapeutic standard concentration of 1250 mg bid.

Treatment Lenalidomide:

Lenalidomide (Revlimid) is a derivative of thalidomide. The exact mechanism of action of these immunomodulatory drugs is not known. Apart from interfering with the immune system, they are also thought to act on angiogenesis. There are multiple mechanisms of action, and they can be simplified by organizing them as mechanisms of action in vitro and in vivo. In vitro, lenalidomide has three main activities: direct anti-tumor effect, inhibition of the micro-environmental support for tumor cells, and an immunomodulatory role. In vivo, lenalidomide induces tumor cell apoptosis directly and indirectly by inhibition of bone marrow stromal cell support, by anti-angiogenic and anti-osteoclastogenic effects, and by immunomodulatory activity. Lenalidomide has a broad range of activities that can be exploited to treat many hematologic and solid cancers.

Lenalidomide is one of the novel drug agents used to treat MM. It is a small molecular analogue of thalidomide that was originally found based on its ability to effectively inhibit tumor necrosis factor alpha (TNF-α) production. Lenalidomide is 50,000 times more potent than thalidomide in inhibiting TNF-α, and has less severe adverse drug reactions.

The most important side effects of lenalidomide are thromboembolism and hematological toxicity. The most common side effects are neutropenia, thrombopenia, anemia, fatigue, constipation, diarrhea, asthenia and rash. In contrast to thalidomide, lenalidomide does not cause neuropathies. Hematotoxicity is dose dependent and easily manageable with dose reductions.

Lenalidomide in combination with dexamethasone is a Swissmedic approved treatment for MM patients who have received at least one prior medicinal therapy. The combination of lenalidomide and dexamethasone compared to dexamethasone alone led to significantly improved progression free survival (median 11.1 vs. 4.6 months) and overall survival (median 38.0 vs. 31.6 months) in patients with relapsed or refractory myeloma in two international phase III trials. More than 1/3 of these patients had previously been treated with the structurally related thalidomide.

Treatment Dexamethasone:

Dexamethasone is a glucocorticosteroid that is used in the treatment of MM, which reduces the activity of the immune system by attaching to receptors in various types of immune cells. In MM, high-dose dexamethasone is used together with chemotherapy to make chemotherapy more effective and to reduce certain side effects of cancer treatment, such as nausea and vomiting.

It appears to cause apoptosis. This means that steroids such as dexamethasone can trigger the destruction of myeloma cells. Typically dexamethasone is given with other agents - such as vincristine, doxorubicin, thalidomide or lenalidomide - to treat MM. It has been found that steroids can increase the ability of chemotherapeutic and immunomodulatory agents such as lenalidomide to destroy myeloma cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have given written informed consent (including the drug-specific informed consent for Revlimid) before registration.
* Multiple myeloma having progressed after at least two months of lenalidomide-containing therapy (progressive disease during treatment with lenalidomide or <60 days after such treatment).
* Measurable disease for myeloma defined as one of the following:

  1. Serum monoclonal protein (M-protein) ≥10 g/L IgG or ≥5 g/L IgA, IgM, IgD
  2. Urine M-protein ≥200 mg/24h
  3. To be considered only if patient has no evidence of measurable disease with one of the criteria above: serum free light chain (FLC) ratio of kappa/lambda either >1.65 or <0.26 (baseline level of involved FLC has to be ≥100 mg/L)
* Adverse events from previous treatment has recovered to grade ≤2.
* Age ≥18 years.
* WHO performance status 0-2.
* Adequate hematological values: neutrophils ≥1 x 109/L, platelets ≥75 x 109/L
* Adequate hepatic function: bilirubin ≤1.5 x ULN, AST and AP ≤2.5 x ULN
* Adequate renal function: calculated creatinine clearance >50 mL/min, according to the formula of Cockcroft-Gault
* Adequate cardiac function: EF ≥40% assessed by echocardiography or MUGA scan
* Negative HIV test.
* Women are not breastfeeding. Women of child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. A negative serum pregnancy test (minimum sensitivity of 25 mIU/ml) before inclusion (within 7 days) into the trial is required for all women of child-bearing potential. Men agree not to father a child during participation in the trial and during 12 months thereafter.
* Patient compliance and geographic proximity allow proper staging and follow-up.

Exclusion Criteria:

* Previous malignancy within 2 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling patient diary, or interfering with compliance for oral drug intake.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy (chemotherapeutical/biological agents, radiation therapy). Treatment in a clinical trial within 30 days prior to trial entry.
* Known hypersensitivity or uncontrolled side effects related to trial drug(s) or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes).
* Unstable cardiovascular disease.
* Known or clinically suspected myeloma manifestations in the central nervous system.
* Previous grade 4 adverse events attributable to treatment with lenalidomide.
* Patients who are on strong CYP3A4 modulators that cannot be replaced at least one week before the first dose of trial drugs and for the period of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose limiting toxicity | Until up to 4 weeks after start of trial therapy
Phase II: Overall response | 16 weeks after the start of trial therapy

SECONDARY OUTCOMES:
Phase I/II: Frequency and percent of occurrence of adverse events during each cycle of treatment, and within patients | Until 30 days after up to 16 weeks of trial therapy
Phase I/II: Disease control, i.e. no progression at 16 weeks after start of trial therapy | At 16 weeks after the start of trial therapy
Phase I/II: Duration of response | Duration from first observation of response to the time of disease progression, with deaths due to causes other than progression censored, assessed until an expected maximum of 3 years
Phase I/II: Overall survival | At 6 months after start of trial therapy
Phase I/II: Progression free survival | Progression free survial time
Phase I/II: Time to progression | Duration from start of treatment to disease progression, with deaths due to causes other than progression censored, assessed until an expected maximum of 3 years
Phase I: Overall response | 16 weeks after the start of trial therapy

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Hitz, MD, Study Chair — Kantonsspital, CH-9007 St. Gallen
Locations (11):
- Italy (2):
  - Istituto Europeo di Oncologia IEO, Milan
  - University of Torino, Torino
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Istituto Oncologico Svizzera Italiana IOSI, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SAKK - SWISS GROUP FOR CLINICAL CANCER RESEARCH — http://sakk.ch/